



### **Consent To Participate In A Research Study**

Group-based mindfulness for patients with chronic low back pain in the primary care setting versus usual care

NCT04129450 PI: Natalia Morone, MD, MS natalia.morone@bmc.org

You are being asked to review this consent addendum because you are participating in a research study at Boston Medical Center entitled "Group-based mindfulness for patients with chronic low back pain in the primary care setting versus usual care".

Please read this consent addendum carefully and take your time making your decision. As your study staff discusses this addendum with you, please ask them to explain any words or information that you do not clearly understand.

You do not have to agree to this addendum to remain in the study.

#### **PURPOSE OF THIS ADDENDUM**

The purpose of this addendum is to request your permission to complete a global mindfulness and life events checklist (LEC-5) scales. These scales include questions that may be sensitive to you, and we understand that it might be difficult for you to answer them. If you feel any emotional discomfort while answering these questions, you are free to stop the questionnaire or skip any of the questions at any time. All the information you provide will be kept confidential and will only be accessible by our study team. We won't reimburse you for completing these questions.

There is no benefit to you from answering these questions. There is a risk of personal discomfort when you disclose personal information. There is a rare risk of breach of confidentiality. This means it is always possible that someone could access the research data and documents and read information about you. The methods we use to protect your confidentiality are described in the main consent.

Except for the activities described in this addendum, the terms of your original consent form remain in full effect.

### QUESTIONS REGARDING THIS ADDENDUM

You should ask the staff members any questions you have about this addendum at any time. Please call us at 617-414-6999 or email us at optimum@bmc.org if you need assistance.

For questions about your rights as a research participant, or to discuss questions, concerns, or suggestions related to the research or this consent addendum, or to obtain information or offer input about the research, please contact the *University of Pittsburgh Human Subjects Protection Advocate toll-free at 866-212-2668*.





# **Consent To Participate In A Research Study**

Group-based mindfulness for patients with chronic low back pain in the primary care setting versus usual care

## **STATEMENT OF CONSENT**

"The purpose of these questionnaires has been explained to me. I have been allowed to ask questions, and my questions have been answered to my satisfaction. I have been told whom to contact if I have questions, to discuss problems, concerns, or suggestions related to the research or this addendum, or to obtain information or offer input about the research. I have read this addendum and agree to the choices I have indicated above, with the understanding that I may withdraw at any time. I provide my verbal consent to complete the scales."